CLINICAL TRIAL: NCT04103476
Title: Atherosclerosis Intervention With Novel Tissue Selective Estrogen Complex Therapy
Brief Title: Advancing Postmenopausal Preventive Therapy
Acronym: APPT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Howard N. Hodis, M.D., Professor of Medicine and Preventive Medicine, Director Atherosclerosis Research Unit, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AG058691 (NIH); R01AG058691 (NIH)
Record Dates: First submitted 2019-09-20; First posted 2019-09-25 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Atherosclerosis; Cognitive Decline
MeSH Terms: conditions — Atherosclerosis; Cognitive Dysfunction | interventions — bazedoxifene; Estrogens, Conjugated (USP)

STUDY DESIGN:
Intervention Model Description: Randomized (1:1), double-blinded, placebo-controlled trial of BZA/CE versus placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization randomly determined with key to treatment groups maintained by a single individual in the data coordinating center (DCC); study product masked with matching placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BZA/CE (Experimental): Oral bazedoxifene 20 mg / conjugated estrogens 0.45 mg
  Interventions: Combination Product: Oral bazedoxifene 20 mg / conjugated estrogens 0.45 mg
- Placebo (Placebo Comparator): Oral matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: Oral bazedoxifene 20 mg / conjugated estrogens 0.45 mg — Oral bazedoxifene 20 mg / conjugated estrogens 0.45 mg
  Arms: BZA/CE
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Advancing Postmenopausal Preventive Therapy (APPT) is a randomized, double-blinded, placebo-controlled trial designed to determine the effects of tissue selective estrogen complex (TSEC) therapy on the progression of subclinical atherosclerosis and cognitive decline in 360 healthy postmenopausal women.

DETAILED DESCRIPTION:
To conduct a double-blinded, placebo-controlled trial to determine the effects of TSEC therapy on the progression of subclinical atherosclerosis in healthy postmenopausal women. A total of 360 postmenopausal women with a uterus who are within 6 years of menopause and 45-59 years of age and without clinical cardiovascular disease and diabetes mellitus will be randomized to Bazedoxifene/Conjugated Equine Estrogen (BZA 20 mg/CE 0.45 mg) or placebo. Recruitment will occur over 3 years and the treatment period will be up to 3 years depending on when an individual is randomized. Rate of change in carotid artery intima-media thickness (CIMT) determined from the distal common carotid artery (CCA) far wall intima-media thickness (IMT) in computer image processed B mode ultrasonograms will be the primary trial endpoint. Arterial stiffness measured from the CCA (same location as CIMT) in computer image processed B mode ultrasonograms will be the secondary trial endpoint. Three composite cognitive measures will be used to test for randomized treatment group differences in cognition; each composite will be considered as co-endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Women with a serum estradiol level <30 pg/ml and cessation of regular menses >6 months who are <6 years postmenopausal and 45-59 years old.

Exclusion Criteria:

* Women with a hysterectomy
* Clinical signs, symptoms or personal history of cardiovascular disease
* Diabetes mellitus or fasting serum glucose >126 mg/dL
* Life threatening illness with prognosis <5 years
* Cirrhosis or liver disease
* History of deep vein thrombosis or pulmonary embolism
* History of breast cancer
* Current use of postmenopausal hormone replacement therapy (HRT) within 1 month of randomization
* Uncontrolled hypertension (>180/>110 mmHg)*
* Plasma triglyceride levels >500 mg/dL
* Serum creatinine >2.0 mg/dL

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 385 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Carotid artery intima-media thickness | At baseline and 6 months, 1 year, 1.5 years, 2 years, 2.5 years and 3 years after randomization
  Rate of change in carotid artery intima-media thickness (CIMT) determined from the distal common carotid artery (CCA) far wall intima-media thickness (IMT) in computer image processed B mode ultrasonograms.

SECONDARY OUTCOMES:
CCA stiffness | At baseline and 6 months, 1 year, 1.5 years, 2 years, 2.5 years and 3 years after randomization
  Arterial stiffness measured from the CCA (same location as CIMT) in computer image processed B mode ultrasonograms.

OTHER OUTCOMES:
Cognitive decline | At baseline and 6 months, 1 year, 1.5 years, 2 years, 2.5 years and 3 years after randomization
  Three composite cognitive measures will be used to test for randomized treatment group differences in cognition; each composite will be considered as co-endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Howard N. Hodis, MD, Principal Investigator — University of Southern California Atherosclerosis Research Unit
Locations (1):
- University of Southern California Atherosclerosis Research Unit, Los Angeles, California, United States